CLINICAL TRIAL: NCT06427928
Title: The Effect of Explaining the Perioperative Process with Our Drawings on Anxiety in Pediatric Patients; Prosperative Randomized Controlled Study
Brief Title: Effect on Anxiety in Pediatric Patients; Successful Randomized Controlled Trial
Acronym: anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Anesthesiology and Reanimation Spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HTSoner
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
Keywords: perioperative anxiety; pediatric; general anhesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Explains the perioperative process with pictures (Active Comparator)
  Interventions: Behavioral: Explains the perioperative process with pictures; Behavioral: The perioperative process is only explained
- The perioperative process is only explained (Other)
  Interventions: Behavioral: Explains the perioperative process with pictures; Behavioral: The perioperative process is only explained

INTERVENTIONS:
Behavioral: Explains the perioperative process with pictures — We will draw pictures of the preoperative area, operating room and postoperative areas of our operating room and explain the process to 34 of the children who will undergo surgery with these pictures. We will explain the process to the other 34 people without the pictures we have. We planned to measure the anxiety levels between the two groups with the modified Yale scale.
Behavioral: The perioperative process is only explained — We will draw pictures of the preoperative area, operating room and postoperative areas of our operating room and explain the process to 34 of the children who will undergo surgery with these pictures. We will explain the process to the other 34 people without the pictures we have. We planned to measure the anxiety levels between the two groups with the modified Yale scale.

SUMMARY:
Preoperative anxiety is characterized by subjective emotions such as irritability, irritability, sadness, and unhappiness. Studies have shown that preoperative anxiety negatively affects children both psychologically and physiologically. Preoperative anxiety occurs in 60-80% of children undergoing anesthesia and surgery and is associated with undesirable consequences such as nightmares, separation anxiety, eating disorders, negative behavioral changes such as increased fear of doctors, increased need for analgesics. The aim of this study is to evaluate the preoperative and pre-sedation anxiety levels in pediatric patients by explaining the peroperative process to the patients with drawings.

ELIGIBILITY:
Inclusion Criteria:

* ASA I patients without any comorbidities who were operated on by the ENT,
* Patients between the ages of 5-12,
* And patients who could be contacted and did not have any anxiety problems were included.

Exclusion Criteria:

* Patients with liver and/or kidney failure, trauma patients, ASAII-III-IV patients, patients with bleeding disorders,
* those using medications that would affect the coagulation system, patients with local anesthetic allergy, patients with immobility and malnutrition, .And patients who did not want to participate in the study were excluded from the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale | surgical ward (T0), in the preoperative waiting area (T1), at the time of separation from the parent to the operating room (T2), upon entry to the operating room (T3), and at the time of starting intravenous induction (T4).
  Activity Interested in his/her surroundings, curious, playing with toys, reading (or other age-appropriate activities); may wander around the waiting room or operating room or go to the parent to retrieve a toy; Can gravitate towards operating room equipment 1
  He is indifferent to his surroundings, does not play, looks at the ground, plays with his hands and fingers, sucks his thumb; may sit very close to the parent while waiting. 2
  Aimless movements directed from the toy towards the parent in an unfocused manner; crazy/exaggerated movements or tricks; writhing, moving on the couch; may push the mask or hug the parent during induction. 3
  The person who actively tries to move away, pushing with his feet and arms, can use his whole body to move away; may not be able to separate from the parent who is running around in the waiting room without focusing, not paying attention to toys, or clinging desperately.4
  Speech Reading (may not speak in relation to the activity), asking

SECONDARY OUTCOMES:
Riker agitation scala | after extubation
  7 -Dangerous Agitation, 6 - Very Agitated, 5 - Agitated, 4 - Calm and Cooperative, 3 - sedated, 2- Very Sedated, 1 -Unarousable
Visual analog scala | surgical ward (T0), in the preoperative waiting area (T1), at the time of separation from their child
  The scale ranged from 0 to 10, where 0 represents not anxious and 10 represents extreme anxiety.
mean arterial pressure | when you come to the operating room table after anesthesia induction Intraoperative 30 minutes after
  mmHg
heart rate | when you come to the operating room table after anesthesia induction Intraoperative 30 minutes after extubation
  beats\minute

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Diyarbakır, Kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No